CLINICAL TRIAL: NCT02856165
Title: High-flow Nasal Oxygen Therapy (Optiflow) in Hospitalized Infant With Moderate-to-severe Bronchiolitis: Multicentric Randomized Controlled Trial
Brief Title: High-flow Nasal Oxygen Therapy in Hospitalized Infant With Moderate-to-severe Bronchiolitis
Acronym: BRONCHOPTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: P150931
Record Dates: First submitted 2016-07-19; First posted 2016-08-04 (Estimated); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Bronchiolitis
Keywords: infant; oxygen therapy; High flow nasal canula oxygen therapy; Bronchiolitis
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High-flow nasal canula oxygen therapy (Experimental): High-flow nasal canula oxygen therapy (HNF) using Optiflow junior system and AIRVO2 turbine (Fisher&Paykel (F&P), NZ)
  Interventions: Device: High-flow nasal canula oxygen therapy
- Low-flow oxygen therapy (Active Comparator): Low-flow oxygen therapy with standard nasal canula
  Interventions: Device: Low-flow oxygen therapy with standard nasal canula

INTERVENTIONS:
Device: High-flow nasal canula oxygen therapy — High-flow nasal canula oxygen therapy (HNF) using Optiflow junior system and AIRVO2 turbine (F&P, NZ) at initial flow to 3l/kg/min (up to a maximum of 20l/min), FiO2 adjusted for SpO2 > 94%.
  Other Names: Optiflow
  Arms: High-flow nasal canula oxygen therapy
Device: Low-flow oxygen therapy with standard nasal canula — flow adjusted to SpO2 > 94% (up to a maximum of 2l/min).
  Other Names: Low-flow oxygen therapy
  Arms: Low-flow oxygen therapy

SUMMARY:
Over the last decade, high-flow nasal oxygen therapy (HFN) has emerged as a new method to provide respiratory support in children with moderate to severe bronchiolitis.

However, any randomized clinical trial (RCT) have demonstrated that earlier support with HFN is superior to standard care including low -flow nasal oxygen therapy to reduce the risk of acute respiratory failure requiring non invasive (or tracheal) ventilation and subsequently the need of PICU transfer.

DETAILED DESCRIPTION:
Open label, non-blinded multi-centre, randomised controlled trial comparing standard care including oxygen delivery via HFN versus standard nasal oxygen therapy in infants admitted to hospital with moderate-to-severe bronchiolitis.

ELIGIBILITY:
Inclusion Criteria:

* first episode of hospitalised bronchiolitis (as defined by American Academy of Pediatrics clinical criterions )
* aged 7 days- 6 months
* transcutaneous SpO2 in room air < 95%
* modified Wood's Clinical Asthma Score (m-WCAS) ≥ 2 et ≤ 5
* agreement of at least one of the parents or legal tutor for his child to participate in biomedical research
* affiliation to social security (beneficiary or entitled), except beneficiary of State medical help

Exclusion Criteria:

* Urgent need for mechanical ventilation support either by nCPAP ou endotracheal route
* Severe form defined by modified Wood's Clinical Asthma Score (mWCAS) exceeding 5 or 6, requiring non invasive ventilation (n CPAP)
* Uncorrected cyanotic heart disease, innate immune deficiency, cranio-facial malformation, congenital stridor, tracheotomy
* Inclusion in other observational study.

Ages: 7 Days to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 268 (Actual)
Dates: Start 2016-10-28 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2017-11-23 (Actual)

PRIMARY OUTCOMES:
patient in treatment failure in each group (control or HFN) requiring non-invasive (or endotracheal) ventilation and ventilation-support free days | Up to an average of 7 days
  Treatment failure is defined if one or more following criteria are met: refractory apnea (> 3/h), oxygen requirement in HFN therapy arm exceeds fraction of inspired oxygen (FiO2) ≥ 40 % or oxygen requirement in standard nasal oxygen therapy arm exceeds >2l/min to maintain oxygen saturation (SpO2) ≥94 %), m-WCAS score increased compared to admission at H6 and/or > 5 , PaCO2 (H6 ) increased compared to admission and > 60-70 mmHg.

SECONDARY OUTCOMES:
Transfer to pediatrics intensive care unit (PICU) | at the end of the follow up (an average of 7 days)
  Numbers of infants transferred to PICU in each arm
Length of stay in paediatric general ward unit | at the end of the follow up (an average of 7 days)
  number of days between the enrolment and return to home or the transfer to PICU when appropriate (treatment failure)
Oxgen-support free days | at the end of the follow up (an average of 7 days)
  number of oxygen support free days
Artificial nutritional-support free days | at the end of the follow up (an average of 7 days)
  number of artificial nutritional-support free days (enteral feeding or intravenous line)
Assessment of short term respiratory status | at the end of the follow up (an average of 7 days)
  Sequential assessment of short term (H1, 6, 12, 24) respiratory status including respiratory rate, heart-rate, SpO2, m-WCAS score, transcutaneous carbon dioxide partial pressure (tcPaCO2).

CONTACTS AND LOCATIONS:
Overall Officials: Philippe DURAND, MD, Principal Investigator — AP-HP, Bicêtre Hospital
Locations (1):
- AP-HP, Bicêtre Hospital, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: Undecided